CLINICAL TRIAL: NCT02005055
Title: Prospective Evaluation of the Use of High-dose-rate Brachytherapy for the Treatment of Recalcitrant Keloids
Brief Title: High Dose Rate Brachytherapy for Treatment of Keloids
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Michiel van Leeuwen, MD, Amsterdam UMC, location VUmc
Other Study IDs: PlastChirVUmc 01
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Keloid
Keywords: Brachytherapy; Radiotherapy; Scar treatment
MeSH Terms: conditions — Keloid | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with recalcitrant keloid scars: All patients with keloids insensitive to other treatments
  Interventions: Procedure: Surgical excision with adjuvant high-dose-rate brachytherapy

INTERVENTIONS:
Procedure: Surgical excision with adjuvant high-dose-rate brachytherapy — The keloid was excised extralesionally and subsequently a metal tipped Varisource catheter was positioned between the dermal edges of the wound, 5 mm below the surface of the skin and extending out of the skin beyond the wound. Primary wound closure was performed and patients were transferred to the radiation department, where the catheter was connected to the Iridium-192 remote control afterloader. The planning target volume was defined as a cylinder along the axis of the scar, with a central diameter of 5mm. Patients received 2 fractions of HighDoseRate brachytherapy. Within 4 hours after the resection, the first brachytherapy fraction of 6 Gy at 5mm of the source axis was given. Within 24 hours after the first fraction a second fraction of 6Gy was administered to a total dose of 12Gy in 2 days. After the second fraction the catheter was gently removed.
  Other Names: Metal tipped Varisource catheter (external diameter: 1.6mm, length: 150cm, Varian medical systems, Palo Alto, USA); Monocryl 4-0 or 5-0; Iridium-192 remote control afterloader (Varisource, Varian medical systems, Palo Alto, USA)

SUMMARY:
This prospective study evaluates the outcome of surgical excision with adjuvant high-dose-rate brachytherapy for the treatment of recalcitrant keloids. Main outcomes are recurrence rate, scar quality and physical complaints.

DETAILED DESCRIPTION:
This prospective evaluation describes the outcome of surgical excision with adjuvant high-dose-rate brachytherapy for the treatment of recalcitrant keloids in a large mixed Fitzpatrick skin type patient population. After intralesional excision, a unique low dose radiation scheme of 2x6Gray (Gy) was administered in 2 fractions: the first within 4 hours, the second within 24 hours. Keloids were evaluated pre- and postoperative (1 week, 3, 6, 12 months, 5years). Scars were measured and recurrence was judged. An evaluation of the outcome of the scars was obtained using the Patient and Observer Scar Assessment Scale. Statistical analyses were conducted using SPSS version 20.0 (SPSS, Inc, Chicago, III)

ELIGIBILITY:
Inclusion Criteria:

* Keloid defined as excessive scar tissue raised above skin level and proliferating beyond the confines of the original lesion. Keloids were distinguished from hypertrophic scars based on the clinical judgment of experienced plastic surgeons and on the age of the scar (>1yr)
* the keloid had been proven insensitive to at least one other treatment
* patients had to be older than 10 years of age.

Exclusion Criteria:

* keloids not suitable for excision with primary closure due to its size or anatomical location
* pregnancy or diabetes

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with recalcitrant keloids meeting inclusion criteria
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Recurrence | At a minimum of one year post surgery
  Recurrence was defined as a growing, pruritic, nodular scar as described by Cosman and Wolff(1)

SECONDARY OUTCOMES:
Scar Quality | Pre- and postoperative
  The scar (pre-operative) and the residual scar (post-operative at 1 week, 3,6,12 months and 5 year) was examined, photographs were taken, surface area was measured and the 'Patient and Observer Scar Assessment Scale' was obtained (2)

CONTACTS AND LOCATIONS:
Overall Officials: Michiel CE Leeuwen van, MD, Principal Investigator — VUmc
Locations (1):
- VUmc, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Cosman B, Wolff M. Bilateral earlobe keloids. Plast Reconstr Surg. 1974 May;53(5):540-3. doi: 10.1097/00006534-197405000-00008. No abstract available. PMID 4821203
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Derived] van Leeuwen MCE, Stokmans SC, Bulstra AJ, Meijer OWM, van Leeuwen PAM, Niessen FB. High-dose-rate brachytherapy for the treatment of recalcitrant keloids: a unique, effective treatment protocol. Plast Reconstr Surg. 2014 Sep;134(3):527-534. doi: 10.1097/PRS.0000000000000415. PMID 25158710
- See also: VU University medical center — http://www.vumc.nl